CLINICAL TRIAL: NCT02968537
Title: Learning to Resist the Urge: Inhibition Training in Abstinent Patients With Alcohol Use Disorders. A Randomized Controlled Trial
Brief Title: Learning to Resist the Urge: Inhibition Training in Abstinent Patients With Alcohol Use Disorders
Acronym: INTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Clinic Südhang (Unknown); Forel Clinic (Other); Psychiatric Center Muensingen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INTRA-2016-00988
Record Dates: First submitted 2016-11-10; First posted 2016-11-18 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Dependence
Keywords: Alcohol use disorders; inhibition; EEG; cortisol; Training; clinical outcome measures
MeSH Terms: conditions — Alcoholism; Inhibition, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Alc-IT (50/50) (morning) (Experimental): Alc-IT (50/50) (morning): This alcohol-specific inhibition-training (Alc-IT) training group will operate with a Go/NoGo ratio of 50/50 (Houben et al. 2011; 2012): This original version of the Alc-inhibition-training will include 80 alcoholic NoGo trials as well as 80 non-alcoholic Go trials. In order to arrive at the same training length while keeping the number of Alc-NoGo-pairings constant and the Go/NoGo-ratio at 50/50, it will additionally include 80 neutral Go-trials as well as 80 neutral NoGo-trials. It will thus consist of 320 trials and take about 10.5 minutes to be completed. In the morning group, this training will be administered within the first 2 hours after awakening.
  Interventions: Behavioral: Alc-IT (50/50) (morning)
- Alc-IT (75/25) (morning) (Experimental): This version of the alcohol-specific inhibition-training (Alc-IT) will operate with a Go/NoGo-ratio of 75/25. It will equally include 80 Alcoholic NoGo-trials and 80 non-alcoholic Go-trials, but now 160 neutral Go-trials will complete the set. This training will also consist of 320 trials and take about 10.5 minutes. In the morning group, this training will be administered within the first 2 hours after awakening.
  Interventions: Behavioral: Alc-IT (75/25) (morning)
- Control-training (morning) (Placebo Comparator): This group will receive an unspecific inhibition training. this training is of the same length and difficulty as the two Alc-inhibition-trainings. In the morning group, this training will be administered within the first 2 hours after awakening.
  Interventions: Behavioral: Control-training (morning)
- Alc-IT (50/50) (afternoon) (Experimental): Alc-IT (50/50) (afternoon): As in the arm "Alc-IT (50/50) (morning)", this alcohol-specific inhibition-training (Alc-IT) group will operate with a Go/NoGo ratio of 50/50 (Houben et al. 2011; 2012): This original version of the Alc-inhibition-training will include 80 alcoholic NoGo trials as well as 80 non-alcoholic Go trials. In order to arrive at the same training length while keeping the number of Alc-NoGo-pairings constant and the Go/NoGo-ratio at 50/50, it will additionally include 80 neutral Go-trials as well as 80 neutral NoGo-trials. It will thus consist of 320 trials and take about 10.5 minutes to be completed. In contrast to the In the morning group, this afternoon group will receive the training in the afternoon.
  Interventions: Behavioral: Alc-IT (50/50) (afternoon)
- Alc-IT (75/25) (afternoon) (Experimental): As in the arm "Alc-IT (75/25) (morning)", this version of the alcohol-specific inhibition-training (Alc-IT) will operate with a Go/NoGo-ratio of 75/25. It will equally include 80 Alcoholic NoGo-trials and 80 non-alcoholic Go-trials, but now 160 neutral Go-trials will complete the set. This training will also consist of 320 trials and take about 10.5 minutes. In contrast to the In the morning group, this afternoon group will receive the training in the afternoon.
  Interventions: Behavioral: Alc-IT (75/25) (afternoon)
- Control-training (afternoon) (Placebo Comparator): As in the arm "Control-training (morning), this group will receive an unspecific inhibition training. This training is of the same length and difficulty as the two Alc-inhibition-trainings. In contrast to the In the morning group, this afternoon group will receive the training in the afternoon.
  Interventions: Behavioral: Control-training (afternoon)

INTERVENTIONS:
Behavioral: Alc-IT (50/50) (morning) — This alcohol-specific inhibition-training (Alc-IT) training group will operate with a Go/NoGo ratio of 50/50 (Houben et al. 2011; 2012): This original version of the Alc-inhibition-training will include 80 alcoholic NoGo trials as well as 80 non-alcoholic Go trials. In order to arrive at the same training length while keeping the number of Alc-NoGo-pairings constant and the Go/NoGo-ratio at 50/50, it will additionally include 80 neutral Go-trials as well as 80 neutral NoGo-trials. It will thus consist of 320 trials and take about 10.5 minutes to be completed. In the morning group, this training will be administered within the first 2 hours after awakening.
  Arms: Alc-IT (50/50) (morning)
Behavioral: Alc-IT (75/25) (morning) — This version of the alcohol-specific inhibition-training (Alc-IT) will operate with a Go/NoGo-ratio of 75/25. It will equally include 80 Alcoholic NoGo-trials and 80 non-alcoholic Go-trials, but now 160 neutral Go-trials will complete the set. This training will also consist of 320 trials and take about 10.5 minutes. In the morning group, this training will be administered within the first 2 hours after awakening.
  Arms: Alc-IT (75/25) (morning)
Behavioral: Control-training (morning) — This group will receive an unspecific inhibition training. this training is of the same length and difficulty as the two Alc-inhibition-trainings. In the morning group, this training will be administered within the first 2 hours after awakening.
  Arms: Control-training (morning)
Behavioral: Alc-IT (50/50) (afternoon) — As in the arm "Alc-IT (50/50) (morning)", this alcohol-specific inhibition-training (Alc-IT) group will operate with a Go/NoGo ratio of 50/50 (Houben et al. 2011; 2012): This original version of the Alc-inhibition-training will include 80 alcoholic NoGo trials as well as 80 non-alcoholic Go trials. In order to arrive at the same training length while keeping the number of Alc-NoGo-pairings constant and the Go/NoGo-ratio at 50/50, it will additionally include 80 neutral Go-trials as well as 80 neutral NoGo-trials. It will thus consist of 320 trials and take about 10.5 minutes to be completed. In contrast to the In the morning group, this afternoon group will receive the training in the afternoon.
  Arms: Alc-IT (50/50) (afternoon)
Behavioral: Alc-IT (75/25) (afternoon) — As in the arm "Alc-IT (75/25) (morning)", this version of the alcohol-specific inhibition-training (Alc-IT) will operate with a Go/NoGo-ratio of 75/25. It will equally include 80 Alcoholic NoGo-trials and 80 non-alcoholic Go-trials, but now 160 neutral Go-trials will complete the set. This training will also consist of 320 trials and take about 10.5 minutes. In contrast to the In the morning group, this afternoon group will receive the training in the afternoon.
  Arms: Alc-IT (75/25) (afternoon)
Behavioral: Control-training (afternoon) — As in the arm "Control-training (morning), this group will receive an unspecific inhibition training. This training is of the same length and difficulty as the two Alc-inhibition-trainings. In contrast to the In the morning group, this afternoon group will receive the training in the afternoon.
  Arms: Control-training (afternoon)

SUMMARY:
The study aims to investigate the effects of a short computerized training as a therapeutic add-on to standard therapy in patients with alcohol-use disorder.

DETAILED DESCRIPTION:
Therapeutic interventions to treat alcohol use disorders (AUD) still need to be improved. A novel alcohol-specific inhibition-training seems to be a promising new intervention. In this study, recently abstinent patients with AUD attending an inpatient treatment program will be randomly assigned to one of two alcohol-specific inhibition-training groups (varying in Go/NoGo-ratio) or to a control condition. Besides the effects on drinking behavior, inhibition and implicit attitudes, the investigators expect the training to influence neurophysiological reactivity to alcohol related stimuli. A subgroup of patients will therefore additionally undergo EEG recording so that the neurophysiological effects of the training can be assessed and related to clinical outcome. Furthermore, since training effects rely on learning processes, the influence of endogenous cortisol level (a consolidation-enhancer which peaks in the morning) on training outcome will be examined by the variation of daytime of the training. All patients' inhibitory control and implicit associations towards alcohol will be measured before and after training. The training effects will be examined on proximal outcome variables (e.g. implicit associations, inhibitory control, abstinence related self-efficacy, craving) and on distal outcome variables at 3-, 6- and 12- months follow-up (e.g. percent abstinent days (primary outcome)).

ELIGIBILITY:
Inclusion Criteria:

* Abstinent patients with an alcohol use disorder in the 12-week inpatient program of the Clinic Südhang or the Forel Clinic,
* Abstained from alcohol for at least 4 weeks (in relation to timepoint when training will start),
* Informed Consent as documented by signature.

Exclusion Criteria:

* Other main psychiatric diagnosis than alcohol use disorder (comorbidity is allowed if the alcohol use disorder is to be considered the main diagnosis),
* other severe substance use disorder (except nicotine), even as secondary diagnosis
* Neurocognitive problems (e.g. Korsakoff syndrome),
* Current medical conditions excluding participation (e.g. acute infectious disease),
* Inability to read and understand the participant's information,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Percent days of abstinence 3-months follow-up. | 3-months follow-up
  Percentage of abstinent days in 3-months follow-up. This will be measured with the timeline follow back (TFB), which is a validated procedure to aid recall of past drinking and evaluates information about drinking behavior.
Inhibition Go/NoGo | Post training, i.e. between 1 and 7 days after completion of the last (i.e. the 6th) training session
  Inhibitory control as assessed with a Go/NoGo task.
Neurophysiology of inhibitory Control (Go/NoGo) | Post training, i.e. between 1 and 7 days after completion of the last (i.e. the 6th) training session
  Neurophysiological correlates of inhibitory control as assessed with EEG-measurement during the Go-NOGo-task. ERPs in response to NoGo-Stimuli will be calculated and the N2/p3-complex will be analyzed
Implicit associations (IAT) | Post training, i.e. between 1 and 7 days after completion of the last (i.e. the 6th) training session
  Implicit associations as assessed with an alcohol-related implicit association task (IAT)
Heavy drinking days in 3 months follow-up | 3 months follow-up
  in 3-months follow-up. This will be measured Heavy drinking days in 3 months follow-up, measured with the timeline follow back (TFB), which is a validated procedure to aid recall of past drinking and evaluates information about drinking behavior.

SECONDARY OUTCOMES:
Abstinence related self-efficacy | Post-training (i.e. between 1 and 7 days after completion of the training session); discharge, 3-, 6- and 12-months follow-up
  Self efficacy will be assessed with the alcohol abstinence self-efficacy scale (AASE).
Craving | Post-training (i.e. between 1 and 7 days after completion of the last training session); discharge, 3-, 6- and 12-months follow-up
  Craving will be measured with the German version of the Obsessive compulsive drinking scale (OCDS-G).
Time to first drink | 3-, 6- and 12-months follow-up
Percent heavy drinking days | 3-, 6- and 12-months follow-up
Inhibition (SST) | Post-training; i.e. between 1 and 7 days after completion of the last (i.e. the 6th) training session
  Inhibitory control will be assessed with a Stop-Signal task

CONTACTS AND LOCATIONS:
Overall Officials: Maria Stein, PhD, Principal Investigator — University of Bern, University Hospital for Psychiatry; Leila Soravia, PhD, Principal Investigator — University of Bern, University Hospital for Psychiatry; Franz Moggi, PD, Principal Investigator — University of Bern, University Hospital for Psychiatry
Locations (3):
- Switzerland (3):
  - Forel Klinik, Ellikon
  - Klinik Südhang, Kirchlindach
  - Psychiatric Center Muensingen, Münsingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tschuemperlin RM, Stein M, Batschelet HM, Moggi F, Soravia LM. Learning to resist the urge: a double-blind, randomized controlled trial investigating alcohol-specific inhibition training in abstinent patients with alcohol use disorder. Trials. 2019 Jul 5;20(1):402. doi: 10.1186/s13063-019-3505-2. PMID 31277683